CLINICAL TRIAL: NCT05368441
Title: Effect of Midazolam Premedication on Mask Ventilation Difficulty During General Anesthesia Induction in Children: A Randomized Clinical Study
Brief Title: Effect of Midazolam Premedication on Mask Ventilation Difficulty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-2021/13
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia Complication
Keywords: premedication; midazolam; anesthesia,general
MeSH Terms: interventions — Midazolam; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The patients will be unaware of the group assignments and monitored in the reception area by a blinded anesthesiologist who will be in charge of the intervention and the evaluation of anxiety and sedation levels.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam-Group M (Experimental): Patients of midazolam group will be treated with midazolam premedication (3 cc mixture of 0.1 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously at waiting area 3 minutes before transportation to an operating room.
  Interventions: Drug: Midazolam
- Control- Group S (Placebo Comparator): Control group patients are treated with 3 cc normal saline at waiting area 3 minutes before transportation to an operating room.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Midazolam — Patients of midazolam group will be treated with midazolam premedication (3 cc mixture of 0.1 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously at waiting area 3 minutes before transportation to an operating room. In anesthesia induction, propofol 2 mg/kg will be given.Before the patients were given muscle relaxants, the patients were evaluated with the Han scale.
  Other Names: Group M
  Arms: Midazolam-Group M
Drug: Saline — Control group patients are treated with 3 cc normal saline at waiting area 3 minutes before transportation to an operating room. In anesthesia induction, propofol 2 mg/kg will be given. Before the patients were given muscle relaxants, the patients were evaluated with the Han's grading scale.
  Other Names: Group S
  Arms: Control- Group S

SUMMARY:
Mask ventilation has great importance during anesthesia induction because it is the only way to oxygenate patients who have lost consciousness and spontaneous breathing. Adequate muscle relaxation and depth of anesthesia may assist with mask ventilation. It is known that premedication to reduce anxiety has a relaxing effect on airway muscles. Midazolam is frequently used in premedication because it has a rapid onset of action and does not cause hemodynamic changes. In addition, midazolam may relax the airway by acting directly on the airway smooth muscle and thus facilitate mask ventilation during anesthesia induction. In this study, we will conduct a randomized controlled trial to evaluate the effect of midazolam premedication on facilitating mask ventilation in children.

DETAILED DESCRIPTION:
American Society of Anesthesiologists (ASA) class I and II patients aged 2-10 years who are scheduled for any elective surgery under general anesthesia will be enrolled. Patients in midazolam group will be treated with midazolam premedication (3 cc mixture of 0.1 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously at waiting area 3 minutes before transportation to an operating room, while 3 cc normal saline will be administered to control group patients. Difficulty of mask ventilation during induction of general anesthesia will be evaluated with the Han Mask Scale. Muscle relaxants will be given for intubation after evaluation. The anxiety and sedation level of patients will be estimated one minute before the intervention and one minute before anesthetic induction in an operating room.

Interventıon descriptıon Patients enrolled in this study are randomly allocated to midazolam group or control group. Total 120 patients will be enrolled. Each group consists of 60 patients. Patients of midazolam group will be treated with midazolam premedication (3 cc mixture of 0.1 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously at waiting area 3 minutes before transportation to an operating room. Control group patients are treated with 3 cc normal saline at waiting area 3 minutes before transportation to an operating room. In anesthesia induction, propofol 2 mg/kg will be given. Before the patients were given muscle relaxants, the patients were evaluated with the Han's mask scale.

ELIGIBILITY:
Inclusion Criteria:

* age 2< and <10 children
* American Society of Anesthesiologists (ASA) class I and II
* Children who are scheduled for any elective surgery under general anesthesia

Exclusion Criteria:

* age <2 or >10 years;
* obesity (body mass index, ≥35 kg/m2);
* craniofacial anomaly;
* allergic reaction to midazolam;
* presence of muscle weakness or dyspnea.
* children posted for any emergency procedure,
* above ASA class II
* children with abnormal airway anatomy,
* children with active respiratory infection in the last 3 weeks,
* children with a past history of chronic respiratory disorder,
* children who are being treated with sedative or anticonvulsive agents

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Difficulty of mask ventilation (Han's grading scale) | At 30 seconds after loss of consciousness
  The Han's scale is a four point grading scale, assigns points based on escalating levels of intervention necessary to ventilate the lungs such as the use of an airway device, two-person ventilation, which are all intended to overcome upper airway resistance to ventilation. (1 point: Easy mask ventilation, 4 point: Impossible - unable to mask ventilate)

SECONDARY OUTCOMES:
Anxiety level, mYPAS (0-100) | One minute before the intervention in waiting area, and one minute before the anesthetic induction in operating room
  The modified Yale Preoperative Anxiety Scale (mYPAS) is an observational measure of children's preoperative anxiety consisting of 27 items divided into 5 categories: Activity, Vocalizations, Emotional Expressivity, State of Arousal and Use of Parent. Scores range from 22.5 to 100 with higher scores indicating greater anxiety.
Sedation level (Modified Observer's assessment of alertness/sedation (MOAA/S) scale) | One minute before the intervention in waiting area, and one minute before the anesthetic induction in operating room
  One minute before the intervention in the waiting area, and one minute before the anesthetic induction in the operating room sedation levels were evaluated with MOAA/S scale. The Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale was developed to measure the level of alertness in subjects who are sedated. The Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scale is frequently used in sedation-related drug and device studies to assess a subject's level of sedation. The MOAA/S ranges from 0 to 5, with a score of 5 defined as awake or minimally sedated, and a score of 0 defined as general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Rafet Yarımoglu, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Yarimoglu R, Basaran B, Et T, Bilge A, Korkusuz M. Midazolam premedication facilitates mask ventilation in children during propofol induction of anesthesia: a randomized clinical trial. BMC Anesthesiol. 2025 Mar 18;25(1):131. doi: 10.1186/s12871-025-03002-4. PMID 40102763